CLINICAL TRIAL: NCT00709449
Title: An Open Study Comparing the Effects of Moxaverine on Ocular Blood Flow in Patients With Age- Related Macular Degeneration, Primary Open Angle Glaucoma and Healthy Control Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Garhöfer, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPHT-011007
Record Dates: First submitted 2008-06-27; First posted 2008-07-03 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Macular Degeneration; Glaucoma; Regional Blood Flow
Keywords: Age-related macular degeneration; Glaucoma
MeSH Terms: conditions — Macular Degeneration; Glaucoma | interventions — moxaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 20 patients with age related macular degeneration
  Interventions: Drug: moxaverine
- 2 (Experimental): 20 patients with primary open angle glaucoma
  Interventions: Drug: moxaverine
- 3 (Experimental): 20 age and sex matched control subjects
  Interventions: Drug: moxaverine

INTERVENTIONS:
Drug: moxaverine — intravenous infusion of 150 mg in 250 ml NaCl, applied over 30 minutes.
  Other Names: Collateral i
  Arms: 1
Drug: moxaverine — intravenous infusion of 150 mg in 250 ml NaCl, applied over 30 minutes.
  Other Names: Collateral i
  Arms: 2
Drug: moxaverine — intravenous infusion of 150 mg in 250 ml NaCl, applied over 30 minutes.
  Other Names: Collateral i
  Arms: 3

SUMMARY:
A number of common eye diseases such as age-related macular degeneration and glaucoma are associated with ocular perfusion abnormalities. Although this is well recognized there is not much possibility to improve blood flow to the posterior pole of the eye in these diseases.

For many years, moxaverine has been used in the therapy of perfusion abnormalities in the brain, the heart and the extremities. This is based on a direct vasodilatatory effect of the drug, but also on the rheological properties of red blood cells. In a recent study the investigators have shown that intravenous moxaverine increases choroidal blood flow in healthy young subjects. The present study aims to investigate, whether moxaverine also improves blood flow in the diseased eye after systemic administration.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 50 years
* Ametropia of less than 6 diopters and anisometropia of less than 2 diopters
* Clear non-lenticular ocular media

AMD patients:

* Patients with nonexudative AMD
* Visual acuity in the study eye > 20/60

Glaucoma patients:

* Unilateral or bilateral primary open angle glaucoma
* At least 3 reliable visual field testings
* Treated intraocular pressure < 21 mmHg,
* Visual field mean deviation MD <10 (Humphrey 30-2)

Healthy control subjects:

* Age- , gender- and sex- matched to the two patient groups,
* Matched with regard to smoking habits of the two patient group
* No observable eye diseases

Exclusion Criteria:

* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of the study drug
* Blood donation during the previous 3 weeks
* Abuse of alcoholic beverages or drugs, participation in a clinical trial in the 3 weeks preceding the study
* Known diabetes mellitus
* Presence of any ocular pathology that interferes with the aims of the present study
* Intraocular surgery within the last 3 weeks
* Hypersensitivity to moxaverine
* Acute gastric bleeding, massive cerebral hemorrhage related to stroke

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Choroidal and optic nerve head blood flow | 2 hours

SECONDARY OUTCOMES:
Retrobulbar flow velocities | 2 hours
Retinal blood flow velocity | 2 hours
Retinal venous and arterial diameters | 2 hours
Intraocular pressure | 2 hours
Systolic and diastolic blood pressure | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria